CLINICAL TRIAL: NCT06672055
Title: A Phase 2b, Double-Blind, Multi-Center, Randomized, Comparator-Controlled Trial to Determine the Relative Efficacy, Safety, and Immunogenicity of the Investigational Oral SARS-CoV-2 Vaccine Tablet Against Currently Approved/Authorized mRNA COVID-19 Injectable Booster Vaccine in Adults Previously Immunized Against COVID-19 Infection
Brief Title: A Study to Evaluate VXA-CoV2-3.3 COVID-19 Vaccine Against Currently Approved/Authorized mRNA COVID-19 Injectable Booster Vaccine in Adults Previously Immunized Against COVID-19 Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: VXA-COV-202
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- VXA-CoV2-3.1 Safety Sentinel Cohort (Experimental): Participants previously immunized against COVID-19 infection will be randomized to receive VXA-CoV2-3.1 (XBB.1.5 vaccine) tablet oral vaccine.
  Interventions: Biological: VXA-CoV2-3.1
- COMIRNATY® Safety Sentinel Cohort (Active Comparator): Participants previously immunized against COVID-19 infection will be randomized to receive COMIRNATY® (variant matched vaccine 2023-2024 formula) injectable COVID-19 vaccine.
  Interventions: Biological: COMIRNATY®
- VXA-CoV2-3.3 (Experimental): If no dose-related toxicities are observed, and upon the recommendation of the Data and Safety Monitoring Board following review of Day 31 safety data in the initial safety cohorts (and possibly immunogenicity data), enrollment will continue with the remaining participants who will be randomized to receive a single dose of VXA-CoV2-3.3 (KP.2 vaccine).
  Interventions: Biological: VXA-CoV2-3.3
- COMIRNATY® (Active Comparator): If no dose-related toxicities are observed, and upon the recommendation of the Data and Safety Monitoring Board following review of Day 31 safety data in the initial safety cohorts (and possibly immunogenicity data), enrollment will continue with the remaining participants who will be randomized to receive a single dose of 2024-2025 formula of COMIRNATY® mRNA COVID-19 injectable vaccine.
  Interventions: Biological: COMIRNATY®

INTERVENTIONS:
Biological: VXA-CoV2-3.1 — Tablets for oral use.
  Arms: VXA-CoV2-3.1 Safety Sentinel Cohort
Biological: COMIRNATY® — Intramuscular (IM) injection.
  Other Names: Pfizer-BioNTech mRNA Vaccine
  Arms: COMIRNATY®; COMIRNATY® Safety Sentinel Cohort
Biological: VXA-CoV2-3.3 — Tablets for oral use.
  Arms: VXA-CoV2-3.3

SUMMARY:
The primary objective of the study is to determine the relative efficacy of the investigational oral severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccine tablet VXA-CoV2-3.3 compared to a currently recommended vaccine for the prevention of symptomatic Coronavirus Disease 2019 (COVID-19).

In order to represent a more recently circulating SARS-CoV-2 variant, the main study endpoints will now evaluate the VXA-CoV2-3.3 (KP.2 strain) vaccine, and not the VXA-CoV2-3.1 (XBB.1.5 strain) vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and above, at time of screening.
2. Completed primary approved/authorized COVID-19 vaccination series with ≥ 2 mRNA vaccine doses.
3. Last COVID-19 vaccine received ≥6 months prior to study vaccination.
4. Male and female participants of childbearing potential must agree to consistently use a highly effective method of contraception from at least 30 days prior to enrollment and through 3 months after the study vaccination.
5. Male participants must refrain from sperm donation from the day of study vaccination through the end of the study. Female participants must refrain from egg donation at least 30 days prior to study vaccination through the end of the study.
6. Is medically stable, as determined by the site investigator (based on review of health status, vital signs, medical history, and physical examination) with screening lab values within normal limits or abnormalities assessed as not clinically significant. Screening platelet count must be >140,000/μL.
7. Agree to not participate in any other SARS-CoV-2 infection prevention trial (vaccine, drug, biologic, PrEP) during participation in the study.
8. Willing and able to provide informed consent prior to initiation of study procedures.
9. Available for all study visits, willing to participate in all study procedures, and not planning to relocate from the area for the duration of the study.
10. Negative rapid molecular Covid test at the screening visit and on Day 1 prior to vaccine dosing.

Exclusion Criteria:

1. Participant has an acute illness as defined by any of the following (note: assessment may be repeated once during screening period) as determined by the site investigator, within 72 hours prior to vaccination as follows:

   1. An acute illness that is nearly resolved, with only minor residual symptoms remaining, is allowable if, in the opinion of the site investigator, the residual symptoms will not interfere with the ability of study staff to assess safety parameters as required by the protocol.
   2. Presence of a fever ≥ 38.0°C (100.4°F) measured orally at baseline, on Day 1 prior to vaccination.
   3. Receipt of antipyretic/analgesic medications within 24 hours prior to vaccine administration.
2. Participant has had a positive COVID test within 90 days prior to screening.
3. Current or planned participation in any other interventional clinical trial.
4. Participation in research involving any investigational product within 45 days prior to study vaccination.
5. Receipt of any approved or authorized products intended to prevent SARS-CoV2 infection within 6 months prior to study vaccination.
6. Receipt or donation of blood products or immunoglobulins within 60 days prior to enrollment or planned administration during the study.
7. Received influenza vaccination within 14 days prior to study vaccination, or any other vaccine within 30 days prior to study vaccination.
8. Any autoimmune or immunodeficiency disease/condition (including and not limited to untreated or advanced HIV infection with CD4 counts <200 cells/mm^3, history of AIDS defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV, severe combined immunodeficiency (SCID), hypogammaglobulinemia, asplenia or functional asplenia).
9. Unstable medical or psychiatric illness (acute or chronic illness) requiring significant medical monitoring and intervention during the 90 days prior to enrollment. Note: diabetes mellitus (Types 1 & 2) are not excluded if assessed by the principal investigator (PI) as well-controlled.
10. Administration of immunosuppressants, systemic glucocorticoids, or other immune-modifying drugs within the following timeframes:

    1. B-cell therapies within the 6 months prior to first study vaccination
    2. Prednisone, ≥20 mg for more than 2 weeks, within the 30 days prior to study vaccination
    3. Other medications in this category, including but not limited to high-dose inhaled corticosteroids (>800 mcg/day of beclomethasone dipropionate or equivalent); antimetabolites; transplant immunosuppressive agents; alkylating agents; cell-depleting agents; or cancer chemotherapeutics, within the 90 days prior to study vaccination.
    4. Any medication for any period of time that, in the opinion of the site investigator, could impede immune response to vaccination.
    5. Use of any dose montelukast OR inhaled, intranasal, intra-articular, or systemic corticosteroids within 2 weeks prior to study vaccination.
    6. Planned use of any of the above medications during the study.
    7. Concomitant allergen immunotherapy (AIT) will be allowed only if the participant is stable in the maintenance phase of AIT. Maintenance AIT should not be dosed for at least 7 days before and 7 days after study vaccine dosing, and the PI must document the treating allergist's approval.
11. Known contraindication to IM injection or blood draws (e.g. bleeding diathesis, acquired coagulopathy, significant bleeding or bruising) or to oral route of administration (unable to swallow tablets).
12. Any known allergies to components contained in the investigational product or comparator or latex allergy (including polyethylene glycol [PEG] allergies) and/or history of serious reactions to vaccination such as anaphylaxis, respiratory problems, hives, or abdominal pain.
13. Women who are pregnant (pregnancy tests will be performed at screening and prior to dosing), breastfeeding, or who plan to become pregnant during the study.
14. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine. Such conditions may include but are not limited to:

    1. Any history of:

       * GI malignancy
       * malabsorption
       * pancreatobiliary disorders
       * inflammatory bowel disease
       * irritable bowel disease
       * hiatal hernia
       * surgical resection
    2. History of diagnosis or treatment in past 5 years of:

       * esophageal or gastric motility disorder
       * gastroesophageal reflux disorder
       * peptic ulcer
       * cholecystectomy.
15. Use of antibiotics, proton pump inhibitors, H2 blockers, or antacids within 7 days prior to study drug administration or planned use from dosing through Day 31.
16. Use of drugs known to affect gastrointestinal motility including glucagon-like peptide 1 (GLP-1) receptor agonists including tirzepatide (Mounjaro) and semaglutide (Wegovy, Ozempic) within 30 days prior to drug administration.
17. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the study.
18. Personal or familial history of hypercoagulable states to include personal past history of deep vein thrombosis (DVT).
19. Personal history of myocarditis or pericarditis.
20. Positive Hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at the screening visit.
21. History of drug, alcohol, or chemical abuse within 1 year of screening.
22. Positive urine drug screen for drugs of abuse at screening (except for occasional marijuana use). Concurrent or planned use of marijuana from dosing through Day 31 is prohibited. Positive urine drug screen (UDS) at screening due to prescribed stimulants will be reviewed on a case by case basis.
23. Cancer, or treatment for cancer, within the past 3 years (excluding fully treated and resolved basal cell carcinoma or squamous cell carcinoma).
24. History of any form of angioedema.
25. History of GI bleeding including hematochezia (blood in stool) or melena (black stool) of unknown etiology or that has not been evaluated.
26. Any history or conditions that may lead to a higher risk of clotting events and/or thrombocytopenia, including:

    1. Familial coagulopathy or personal history of bleeding disorder or thrombosis
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments
    3. History of autoimmune or inflammatory disease
    4. Presence of any of the following conditions known to increase the risk of thrombosis within 6 months prior to screening:

       * Recent surgery other than fully healed cesarean delivery or excision/ biopsy of cutaneous lesions
       * Immobility (confined to bed or wheelchair for 3 or more successive days)
       * Head trauma with loss of consciousness or documented brain injury
       * Receipt of anticoagulants for prophylaxis of thrombosis
       * Recent clinically significant infection including hospitalization for COVID-19 related illness.
27. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the investigational product or interpretation of study results.
28. Study team member or first-degree relative of any study team member (inclusive of sponsor and site personnel involved in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10400 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
KP.2 Cohorts: Percentage of Participants with First Occurrence of Symptomatic Polymerase Chain Reaction (PCR)-Positive COVID-19 at 14 Days Post-vaccination | Up to approximately Day 14
KP.2 Cohorts: Percentage of Participants with First Occurrence of Symptomatic PCR-Positive COVID-19 at 12 Months Post-vaccination | Up to approximately 12 months
XBB Sentinel Cohorts: Percentage of Participants who Experience any Solicited Local Reactogenicity Through 7 Days Post-vaccination | Up to approximately Day 7
XBB Sentinel Cohorts: Percentage of Participants who Experience any Solicited Systemic Reactogenicity Through 7 Days Post-vaccination | Up to approximately Day 7
XBB Sentinel Cohorts: Percentage of Participants who Experience Unsolicited Adverse Events (AEs) Through 30 Days Post-vaccination | Up to approximately Day 30
XBB Sentinel Cohorts: Percentage of Participants who Experience Treatment-emergent Adverse Events (TEAEs) Through 12 Months Post-vaccination | Up to approximately 12 months
  An AE is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. An AE of special interest (AESI) is an AE (serious or non-serious) of scientific and medical concern specific to the sponsor's product or program. Medically attended AEs (MAAEs) are defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic. A serious TEAE (SAE) is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
XBB Sentinel Cohorts: Percentage of Participants With any Clinically Significant Abnormal Safety Laboratory Results Within 7 Days Pots-vaccination | Up to approximately Day 7

SECONDARY OUTCOMES:
KP.2 Cohorts: Percentage of Participants with First Occurrence of Symptomatic PCR-Positive COVID-19 Within 14 Days and 12 Months Post-vaccination in Participants with Specified Body Mass Index (BMI) | Up to approximately 12 months
KP.2 Cohorts: Percentage of Participants with First Occurrence of Symptomatic PCR-Positive COVID-19 within 0 and 6 Months Post-vaccination | Up to approximately 6 months
KP.2 Cohorts: Percentage of Participants with First Occurrence of Symptomatic PCR-Positive COVID-19 within 6 and 12 Months Post-vaccination | Up to approximately 12 months
KP.2 Cohorts: Number of Participants with First Occurrence of Asymptomatic PCR-Positive COVID-19 within 14 Days and 12 Months Post-vaccination | Up to approximately 12 months
KP.2 Cohorts: Number of Participants with First Occurrence of Severe PCR-Positive COVID-19 within 14 Days and 12 Months Post-vaccination | Up to approximately 12 months
KP.2 Cohorts: Percentage of Participants who Experience any Solicited Local Reactogenicity Through 7 Days Post-vaccination | Up to approximately Day 7
KP.2 Cohorts: Percentage of Participants who Experience any Solicited Systemic Reactogenicity Through 7 Days Post-vaccination | Up to approximately Day 7
KP.2 Cohorts: Percentage of Participants who Experience Unsolicited AEs Through 30 Days Post-vaccination | Up to approximately Day 30
KP.2 Cohorts: Percentage of Participants who Experience TEAEs Through 12 Months Post-vaccination | Up to approximately 12 months
  An AE is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurred after the participant received study treatment. An AESI is an AE (serious or non-serious) of scientific and medical concern specific to the sponsor's product or program. MAAEs are defined as AEs with medically attended visits including hospital, emergency room, urgent care clinic. An SAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
KP.2 Cohorts: Percentage of Participants With any Clinically Significant Abnormal Safety Laboratory Results Within 7 Days Pots-vaccination | Up to approximately Day 7
KP.2 Cohorts: Concentration of SARS-CoV-2 Specific Serum Neutralizing Antibodies (nAb) Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Fold Rise of SARS-CoV-2 Specific Serum nAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Concentration of Serum Immunoglobulin G (IgG) Binding Antibody (bAb) Against Spike Protein (S) and Receptor Binding Domain (RBD) Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Fold Rise of Serum IgG Anti-S or RBD Specific bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Concentration of Serum Immunoglobulin A (IgA) bAb Against S and RBD Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Fold Rise of Serum IgA Anti-S or RBD Specific bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Concentration of S and RBD-specific Saliva IgA bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Fold Rise of S and RBD-specific Saliva IgA bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Concentration of S and RBD-specific Nasal Lining Fluid (NLF) IgA bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Fold Rise of S and RBD-specific NLF IgA bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Percentage of Participants With 2, 3, and 4 Fold Rise in S or RBD-Specific Serum IgG and IgA bAb, Serum nAb, Saliva IgA bAb, and NLF IgA bAb Post-vaccination | Day 1 and Months 1, 3, 6, and 12
KP.2 Cohorts: Concentration of Intracellular T Cell Cytokine and Cell Surface Marker at Day 1 and 1 Month Post-vaccination | Day 1 and Month 1
KP.2 Cohorts: Concentration of Intracellular T Cell Cytokine and Cell Surface Marker at 3, 6, and 12 Months Post-vaccination | Months 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (145):
- United States (145):
  - Pinnacle Research Group, Anniston, Alabama
  - Core Clinical Trials - Central Alabama Research LLC, Birmingham, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Avacare - Lenzmeier Family Medicine, Glendale, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Velocity Clinical Research - MedPharmics - Phoenix, Phoenix, Arizona
  - Foothills Research Center, Phoenix, Arizona
  - Avacare (CCT) - Fiel Family & Sports Medicine, Tempe, Arizona
  - Baptist Health Center for Clinical Research - Little Rock, Little Rock, Arkansas
  - Elligo Health Research (BTC/ClinEdge) - Core Healthcare Group, Cerritos, California
  - Velocity Clinical Research - Chula Vista (eStudySite - Chula Vista), Chula Vista, California
  - Avacare - Benchmark Research - SOCAL-Colton, Colton, California
  - Altasciences Los Angeles (Formerly WCCT Global), Cypress, California
  - Ark Clinical Research - Fountain Valley, CA, Fountain Valley, California
  - Velocity Clinical Research - San Diego (eStudySite - La Mesa), La Mesa, California
  - Ark Clinical Research - Long Beach, CA, Long Beach, California
  - Velocity Clinical Research (National Research Institute) - Panorama City, Los Angeles, California
  - Northern California Research, Sacramento, California
  - Avacare - Benchmark Research - Sacramento, Sacramento, California
  - Velocity Clinical Research - Gardena, Santa Ana, California
  - Elite Research Network (ERN) - Legacy Clinical Trials, Colorado Springs, Colorado
  - Tekton Research - Fort Collins, Fort Collins, Colorado
  - Avacare - Critical Care, Pulmonary and Sleep Associates, Lakewood, Colorado
  - Tekton Research - Colorado - Longmont, Longmont, Colorado
  - Paradigm Clinical Research - Wheat Ridge, Wheat Ridge, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Chase Medical Research, Waterbury, Connecticut
  - Velocity Clinical Research - Washington DC, Washington D.C., District of Columbia
  - AMR - Miami (Clinical Research of South Florida), Coral Gables, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Velocity Clinical Research - New Smyrna Beach, Edgewater, Florida
  - Fleming Island Center For Clinical Research, Fleming Island, Florida
  - AMR - Fort Myers - Clinical Physiology Associates, Fort Myers, Florida
  - Velocity Clinical Research - Hallandale Beach (MD Clinical), Hallandale, Florida
  - ENCORE - Nature Coast Clinical Research Inverness, Inverness, Florida
  - ENCORE - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Headlands Research - JEM Research - Lake Worth, Lake Worth, Florida
  - Accel Research Sites - Lakeland, Lakeland, Florida
  - Accel Research Sites (ARS) - St. Petersburg - Largo, Largo, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - SRA Trials LLC - Miami Clinical Trials at Suncoast Research Associates, Miami, Florida
  - Atlas Clinical Research - Suncoast Clinical Research - Pasco County, New Port Richey, Florida
  - Biscayne Clinical Research, North Miami Beach, Florida
  - K2 Medical Research - South Orlando, Orlando, Florida
  - Boca Raton Clinical Research (BRCR) Global - Weston, Plantation, Florida
  - ENCORE - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - IMA Clinical Research - St. Petersburg, St. Petersburg, Florida
  - hyperCORE - Centricity Research Columbus, Columbus, Georgia
  - Javara Research - Privia Medical Group Georgia, Fayetteville, Georgia
  - Privia Health - SouthCoast Health, Fayetteville, Georgia
  - Avacare (CCT) - Lifeline Primary Care, Lilburn, Georgia
  - hyperCORE - Centricity Research (IACT Health) - Rincon, Rincon, Georgia
  - Velocity Clinical Research - Savannah, Savannah, Georgia
  - Velocity Clinical Research - Boise (Meridian), Meridian, Idaho
  - IMA Clinical Research - Chicago, Chicago, Illinois
  - Accellacare - Duly Health and Care, Lombard, Illinois
  - Velocity Clinical Research - Valparaiso (Buynak Clinical Research), Valparaiso, Indiana
  - Accellacare - McFarland Clinic, Ames, Iowa
  - Velocity (Meridian) Clinical Research - Sioux City, Sioux City, Iowa
  - AMR - El Dorado - Heartland Research Associates, El Dorado, Kansas
  - Johnson County Clin-Trials, Lenexa, Kansas
  - AMR - Newton (Heartland Research Associates), Newton, Kansas
  - AMR - Wichita West - Heartland Research Associates, Wichita, Kansas
  - AMR - Wichita East - Heartland Research Associates, Wichita, Kansas
  - AMR - Lexington (Central Kentucky Research Associates), Lexington, Kentucky
  - Velocity (Meridian) Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Avacare - Benchmark Research - New Orleans-North Shore, Covington, Louisiana
  - Velocity Clinical Research - MedPharmics - Covington, Covington, Louisiana
  - Boca Raton Clinical Research (BRCR) Global USA - New Orleans, Gretna, Louisiana
  - Velocity Clinical Research - MedPharmics - Lafayette, Lafayette, Louisiana
  - Avacare - Benchmark Research - Metairie, Metairie, Louisiana
  - AMR - New Orleans - Center for Clinical Research, New Orleans, Louisiana
  - Javara Research - Privia Medical Group Mid-Atlantic - Annapolis, Annapolis, Maryland
  - Pharmaron, Baltimore, Maryland
  - Avacare (CCT) - Advanced Primary and Geriatric Care, Rockville, Maryland
  - Velocity (Meridian) Clinical Research - Rockville, Rockville, Maryland
  - Javara Research - Mankato Clinic, Mankato, Minnesota
  - Velocity Clinical Research - MedPharmics - Gulfport, Gulfport, Mississippi
  - Avacare (CCT) - Clay Platte Family Medicine Clinic, Kansas City, Missouri
  - Avacare (CCT) - Skyline Medical Center, Elkhorn, Nebraska
  - Velocity (Meridian) Clinical Research - Grand Island, Grand Island, Nebraska
  - Be Well Clinical Studies - Nebraska, Lincoln, Nebraska
  - Velocity (Meridian) Clinical Research - Omaha, Omaha, Nebraska
  - hyperCORE - ActivMed Practices and Research - Portsmouth, Portsmouth, New Hampshire
  - DM Clinical Research - Jersey City, Jersey City, New Jersey
  - Velocity Clinical Research - Alburquerque, Albuquerque, New Mexico
  - AXCES Research & Health - Santa Fe, Santa Fe, New Mexico
  - IMA Clinical Research - Albany, Suite 202, Albany, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - IMA Clinical Research - Manhattan, New York, New York
  - Atlas Clinical Research - Rochester Clinical Research, Rochester, New York
  - Cary Medical Group, Cary, North Carolina
  - Velocity Clinical Research - Durham, Durham, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare - Rocky Mount, Rocky Mount, North Carolina
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accellacare - Piedmont Healthcare, Statesville, North Carolina
  - Accellacare - Tradd Court, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland (Rapid Medical Research), Beachwood, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati (New Horizons Clinical Research - Blue Ash), Cincinnati, Ohio
  - Tekton Research - Oklahoma - Magnolia Court, Moore, Oklahoma
  - Tekton Research - Delaware Pointe, Tulsa, Oklahoma
  - Tekton Research - Oklahoma - Primary Health Partners, Yukon, Oklahoma
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Avacare (CCT) - Hatboro Medical Associates, Hatboro, Pennsylvania
  - Atlas Clinical Research - Suburban Research Associates - Media Office, Media, Pennsylvania
  - Velocity Clinical Research - Providence (East Greenwich), East Greenwich, Rhode Island
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - Velocity Clinical Research - Charleston, Charleston, South Carolina
  - Velocity Clinical Research - Columbia (VitaLink), Columbia, South Carolina
  - Accellacare - Charleston, Mt. Pleasant, South Carolina
  - Trial Management Associates - Myrtle Beach, Myrtle Beach, South Carolina
  - hyperCORE International - Coastal Carolina Research Center, North Charleston, South Carolina
  - Velocity Clinical Research - Union (Vitalink), Union, South Carolina
  - Accellacare - PMG Research of Bristol, Bristol, Tennessee
  - Alliance for Multispecialty Research (AMR) - Corporate, Knoxville, Tennessee
  - Accellacare of Knoxville, Knoxville, Tennessee
  - Velocity Clinical Research - Abilene, Abilene, Texas
  - IMA Clinical Research - Austin, Austin, Texas
  - Tekton Research - Austin, Austin, Texas
  - Orion Clinical Research, Austin, Texas
  - Velocity Clinical Research - Austin, Austin, Texas
  - Tekton Research - Beaumont, Beaumont, Texas
  - PanAmerican Clinical Research - Brownsville, Levee Street, Brownsville, Texas
  - Cedar Health Research - Arlington/Euless, Euless, Texas
  - EmVenio Research - Fort Worth, TX, Fort Worth, Texas
  - Avacare - Benchmark Research Fort Worth, Fort Worth, Texas
  - DM Clinical Research - CyFair Clinical Research Center, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - DM Clinical Research - Tomball - Multiple Specialties, Tomball, Texas
  - Velocity Clinical Research - Waco (formerly: Impact Research Institute), Waco, Texas
  - Avacare (CCT) - Ogden Clinic - Grand View, Roy, Utah
  - Avacare (CCT) - Olympus Family Medicine, Salt Lake City, Utah
  - South Ogden Family Medicine, South Ogden, Utah
  - Health Research of Hampton Roads, Newport News, Virginia
  - AMR - Norfolk (Clinical Research Associates of Tidewater), Norfolk, Virginia
  - Centricity Research (IACT Health) - Suffolk Primary Care, Suffolk, Virginia
  - Velocity Clinical Research - Medford, Spokane, Washington
  - Velocity Clinical Research - Spokane, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No